CLINICAL TRIAL: NCT01455974
Title: The Effects of Lowering Dialysate Sodium in Hypertensive Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Yi-Lun Zhou, Associate professor, Capital Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2011-09-28; First posted 2011-10-20 (Estimated); Last update posted 2011-10-20 (Estimated); Status verified 2011-10

CONDITIONS: Hypertension; Arteriosclerosis; Left Ventricular Hypertrophy
Keywords: hypertension; arterial stiffness; left ventricular hypertrophy
MeSH Terms: conditions — Hypertension; Arteriosclerosis; Hypertrophy, Left Ventricular

ARMS (1):
- Dialysate sodium set at 136 mmol/L (Experimental)
  Interventions: Other: Decreasing dialysate sodium from 138 mmol/L to 136 mmol/L

INTERVENTIONS:
Other: Decreasing dialysate sodium from 138 mmol/L to 136 mmol/L — After 1-month period of dialysis with standard dialysate sodium concentration 138mmol/L, patients were followed up over a 1-year period with dialysate sodium set at 136mmol/L, without changes in instructions to patients about dietary sodium.

SUMMARY:
Unfavorably high sodium intakes remain prevalent around the world. A negative sodium gradient in hemodialysis treatment results in absolute sodium removal via diffusive transport of sodium from the blood to the dialysate, and it may be a potentially useful tool to improve sodium loading due to excess dietary sodium intake.

The purpose of this study is to determine whether a in small negative sodium gradient could improve blood pressure level, arterial stiffness and left ventricular hypertrophy in hypertensive hemodialysis patients, who had been achieving and maintaining their dry weight assessed by bioimpedance spectroscopy.

DETAILED DESCRIPTION:
A number of studies have shown that lowering dialysate sodium concentration could improve blood pressure (BP) control, and the lower BPs are considered to be a result of an improvement in volume status via increasing sodium removal. However, sodium, apart from volume, may have an independent effect on BP regulation. It is speculated that a reduction in exchangeable sodium, even without a change in body water content, may improve BP control. Unfortunately, as of yet, no clinical studies have actually provided the evidence in this field.

In general population, dietary salt loading produces significant increase in aortic pulse wave velocity, which is reversed by lowering sodium intake. To the investigators knowledge, the effect of sodium on arterial stiffness has not been investigated in hemodialysis patients.

A regression of left ventricular hypertrophy (LVH) has been achieved through strict dietary sodium restriction in hemodialysis patients. Lack of effect on LVH was observed in low sodium dialysis which may be due to the shorter time interval.

ELIGIBILITY:
Inclusion Criteria:

* They had been on HD for more than 1 year.
* They had had no clinical cardiovascular disease during 3 months preceding entry into the study, with left ventricular ejection fraction over 40%.
* Their residual daily urine output was lower than 100 ml/day.
* They had achieved their dry weight assessed by bioimpedance technique and clinical examination for at least 3 months.
* A mean interdialytic ambulatory BP of >135/85 mmHg.
* Averaging the last six available monthly pre-dialysis plasma sodium concentrations over the preceding 12 months >138mmol/l.

Exclusion Criteria:

* They had known acute inflammatory event, malignant disease, and the serum albumine<30g/l.
* They were diabetic and hypotension prone.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-10; Primary Completion 2011-02 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Changes in 44-hour ambulatory systolic and diastolic blood pressure | Baseline, 4 months, and 12 months
  The change is calculated as the 4 months minus baseline, and the 12 months minus baseline

SECONDARY OUTCOMES:
Changes in aortic pulse wave velocity and left ventricular mass index | Baseline, 4 months, and 12 months
  The change is calculated as the 4 months minus baseline, and the 12 months minus baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nephrology, Chao-Yang Hospital, Capital Medical University, Beijing, China